CLINICAL TRIAL: NCT06525519
Title: Dose Study of Anti-T Lymphocyte Globulin (ATLG) in GVHD Prophylaxis
Brief Title: Comparison of Different Dose of Anti-T Lymphocyte Globulin (ATLG) in Haploidentical HSCT for GVHD Prophylaxis
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024027
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-06

CONDITIONS: Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATLG-20 mg/kg (Experimental): ATLG 20mg/kg group refers to treatment with ATLG in the total dose of 20mg/kg.
  Interventions: Drug: ATLG
- ATLG-30mg/kg (Experimental): ATLG 30mg/kg group refers to treatment with ATLG in the total dose of 30mg/kg.
  Interventions: Drug: ATLG

INTERVENTIONS:
Drug: ATLG — 5 mg/kg/day IV for 4 consecutive days (day-5 to -2 before transplantation). All transplant recipients will receive myeloablative conditioning or modified myoloablative conditioning and standard GVHD prophylaxis.
  Arms: ATLG-20 mg/kg
Drug: ATLG — 7.5mg/kg/day IV for 4 consecutive days (day-5 to -2 before transplantation). All transplant recipients will receive myeloablative conditioning or modified myoloablative conditioning and standard GVHD prophylaxis.
  Arms: ATLG-30mg/kg

SUMMARY:
This study aims to compare the incidence of graft-versus-host disease (GVHD) in haploidentical hematopoietic stem cell transplant recipients who receive varying doses of anti-T lymphocyte globulin (ATLG) for GVHD prophylaxis. Our primary objective is to determine the optimal dose of ATLG for preventing acute GVHD (aGVHD). Additionally, we plan to evaluate the impact of different doses of ATLG on post-transplant viral infections and other clinical outcomes.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is the only therapeutic option for many hematological malignancies. Haploidentical related donor transplantation is now considered an important allo-HSCT. GVHD prevention has a crucial role in post-transplant outcomes by potentially interfering with the graft-versus-leukemia (GVL) effect and immune reconstitution. In vivo T cell depletion (TCD) modalities, including anti-T lymphocyte globulin (ATLG)-based protocols have been widely used worldwide for GVHD prophylaxis.

Several European studies have shown that a dose of 30mg/kg of ATLG can effectively prevent GVHD with acceptable safety. But, the most commonly reported dose among Chinese population is 20mg/kg. Additionally, the main type of allo-HSCT in China is haploidentical transplantation. The application experience of ATLG in Europe mainly focuses on sibling and unrelated donor transplants. There is still a lack of sufficient exploration on the optimal dose of ATLG in GVHD prevention in haploidentical transplantation.

In this prospective multiple-center randomized trial, we aim to compare the effects of different doses of ATLG on GVHD prevention, risk of viral infection, and patient survival after haploidentical transplantation.

ELIGIBILITY:
Inclusion Criteria:

* 1，Age ≥ 16 and ≤ 65 years 2, Patients undergoing Haplo-identical hematopoietic stem cell transplantation 3, AML and ALL in complete cytologic response or MDS requiring allogeneic stem cell transplantation 4, ECOG performance status ≤ 2

Exclusion Criteria:

* 1，Pregnant or lactating females 2，Patients who have previously undergone allogeneic hematopoietic stem cell transplantation or organ transplantation 3, Patients with major organ abnormal including renal, liver, lung , heart and/or CNS diseases, where these diseases or others cannot be controlled by treatment and may affect the completion of this study 4, Uncontrolled infection 5, Seropositivity for HIV or HTLV-1 or active hepatitis B or C 6, Patients with any other complications that may affect this study or with a history of malignant diseases.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade II-IV acute Graft Versus Host Disease (GVHD) | At day 100 post-transplantation
  aGVHD was graded according to standard criteria

SECONDARY OUTCOMES:
Incidence of moderate to severe chronic GVHD (cGVHD) | 1 year
  Chronic GVHD was assessed in patients alive after day 100. cGVHD was graded according to standard criteria.
Incidence of Epstein-Barr virus(EBV) viremia | 180 days
  Incidence of EBV viremia within 180 days
Survival without relapse and moderate to severe GVHD | 1 year
  Rate of patients remain alive without disease relapse or progression (bone marrow blast >5% or extra medullary diseases) and without documentation of grade III-IV acute GVHD and moderate to severe chronic GVHD

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The Southwest Hospital of Amu, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Bethune Hospital of Jilin University, Jilin, Jilin
  - Tai'an City Central Hospital, Taian, Shandong
  - People's Liberation Army The General Hospital of Western Theater Command, Chengdu, Sichuan